CLINICAL TRIAL: NCT03859271
Title: Using Information Communication Technology to Deliver Brief Motivational Interviewing to Promote Regular Physical Activity Among Chinese Childhood Cancer Survivors: A Randomized Controlled Trial
Brief Title: Using Information Communication Technology to Deliver Brief Motivational Interviewing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: UW 19-053
Record Dates: First submitted 2019-02-27; First posted 2019-03-01 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2020-11

CONDITIONS: Childhood Cancer
Keywords: Physical activity
MeSH Terms: conditions — Neoplasms; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- brief motivational interviewing (Experimental): Participants will receive BMI and instant messaging delivered by a trained research nurse. At the time of recruitment, both children and parents will receive an education talk on the significance of and misconceptions about regular physical activity for cancer survivors and strategies for overcoming barriers to engaging in physical activity. Parents will then receive a face-to-face BMI to motivate their children to engage in regular physical activity. Parents will also be encouraged to motivate their children to intensify their physical activity levels progressively, with the ultimate goal of achieving the Global Recommendations on Physical Activity on Health suggested by the World Health Organization. Additionally, they will be invited to download a mobile health application from the Centre for Health Protection, Department of Health, HKSAR website that contains information on physical activity.
  Interventions: Behavioral: Brief motivational interviewing
- Placebo Control (Placebo Comparator): Children and parents will receive the education talk on physical activity and ask to download the mobile health application that contains information on physical activity at the time of recruitment similar to the intervention group. However, parents will not receive BMI and instant messaging throughout the study period.
  Interventions: Behavioral: Placebo control

INTERVENTIONS:
Behavioral: Brief motivational interviewing — Children and parents will receive BMI and instant messaging delivered by a trained research nurse. At the time of recruitment, both children and parents will receive an education talk on the significance of and misconceptions about regular physical activity for cancer survivors and strategies for overcoming barriers to engaging in physical activity. Parents will then receive a face-to-face BMI to motivate their children to engage in regular physical activity. Parents will also be encouraged to motivate their children to intensify their physical activity levels progressively, with the ultimate goal of achieving the Global Recommendations on Physical Activity on Health suggested by the World Health Organization. Additionally, they will be invited to download a mobile health application from the Centre for Health Protection, Department of Health, HKSAR website that contains information on physical activity.
  Arms: brief motivational interviewing
Behavioral: Placebo control — Children and parents will receive the education talk on physical activity and ask to download the mobile health application that contains information on physical activity at the time of recruitment similar to the intervention group. However, parents will not receive BMI and instant messaging throughout the study period.
  Arms: Placebo Control

SUMMARY:
This study aims to examine the efficacy of using Information Communication Technology (ICT) to deliver brief Motivational Interviewing (BMI) to promote regular physical activity among Hong Kong Chinese childhood cancer survivors.

DETAILED DESCRIPTION:
A substantial body of evidence has indicated that improved childhood cancer survival has inevitably been accompanied by increased chronic physical problems and adverse psychological late-effects of cancer and its treatment. The frequently reported physiological and psychological sequelae included cancer-related fatigue, reduced muscle strength, decreases in functional capacity, activity intolerance, depression and distorted self-esteem, which in turn severely comprises their quality of life.

There is a growing body of evidence highlighting the beneficial effects of physical activity on the physiological and psychological health of childhood cancer survivors. Particularly, substantial evidence reveals that engaging in regular moderate-intensity physical activity can help ameliorate some of the treatment-related adverse effects experienced by childhood cancer survivors, such as reduce cancer-related fatigue, enhance muscle strength, improve cardiovascular fitness and eventually lead to a better quality of life.

Evidence demonstrates that education alone is insufficient or unlikely to change behavior. Motivational interviewing (MI) is a directive, client-centered counseling strategy which differs from prevailing patient education to support clients to explore and resolve their ambivalence about changing their behaviors. Meanwhile, there is an increase in the use of Information Communication Technology (ICT) for health care delivery and health promotion. Using instant messaging (i.e. WhatsApp or WeChat) allows quick, direct and continuing professional advice and support for the parents to promote their child's level of physical activity. Therefore, the aim of this study is to examine the efficacy of using ICT to deliver BMI to promote regular physical activity among Hong Kong Chinese childhood cancer survivors.

ELIGIBILITY:
The Inclusion Criteria for eligible Hong Kong Chinese childhood cancer survivals are as follows:

* Aged 9 to 16 years;
* Able to speak Cantonese and read Chinese;
* Had completed cancer treatment at least six months previously; and
* currently do not engage in regular physical exercise.

Exclusion Criteria:

* The investigators will exclude childhood cancer survivors with evidence of recurrence or second malignancies, and those with physical impairment or cognitive and learning problems identified from their medical records.

Additionally, parents (either father or mother; the primary caregiver of childhood cancer survivors) must be able to:

* Speak Cantonese and read Chinese,
* Use a smartphone and can use an instant messaging tool (e.g., WhatsApp/WeChat); and
* Are willing to receive health promotion advice and interact with our interventionist via WhatsApp/WeChat on a smartphone throughout the study period.

Ages: 9 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 161 (Actual)
Dates: Start 2019-03-11 (Actual); Primary Completion 2021-01-29 (Actual); Study Completion 2021-01-29 (Actual)

PRIMARY OUTCOMES:
Change in levels of physical activity from baseline to 12-month follow-up between intervention and control group | 12-month follow-up
  The primary outcome measure is the physical activity levels of subjects at 12-month follow-up when compare to baseline. The Chinese University of Hong Kong: Physical Activity Rating for Children and Youth (CUHK-PARCY) will be used to assess participants' physical activity levels. It is a one-item scale, scores ranging from 0-2, 3-6 and 7-10 indicate low, moderate and high levels of physical activity respectively.

SECONDARY OUTCOMES:
Levels of physical activity at baseline | baseline
  The Chinese University of Hong Kong: Physical Activity Rating for Children and Youth (CUHK-PARCY) will be used to assess participants' physical activity levels. It is a one-item scale, scores ranging from 0-2, 3-6 and 7-10 indicate low, moderate and high levels of physical activity respectively.
Change in levels of physical activity from baseline at 1-month follow-up between intervention and control group | 1-month follow-up
  The Chinese University of Hong Kong: Physical Activity Rating for Children and Youth (CUHK-PARCY) will be used to assess participants' physical activity levels. It is a one-item scale, scores ranging from 0-2, 3-6 and 7-10 indicate low, moderate and high levels of physical activity respectively.
Change in levels of physical activity from baseline at 3-month follow-up between intervention and control group | 3-month follow-up
  The Chinese University of Hong Kong: Physical Activity Rating for Children and Youth (CUHK-PARCY) will be used to assess participants' physical activity levels. It is a one-item scale, scores ranging from 0-2, 3-6 and 7-10 indicate low, moderate and high levels of physical activity respectively.
Change in levels of physical activity from baseline at 6-month follow-up between intervention and control group | 6-month follow-up
  The Fatigue Scale - Child will be used to assess the fatigue of subjects who are 7 to 12 years old. For those aged 13 to 18, their fatigue levels will be measured by the Fatigue Scale - Adolescent.
Levels of cancer-related fatigue at baseline | Baseline
  The Fatigue Scale - Child will be used to assess the fatigue of subjects who are 7 to 12 years old. It contains 13 items, rated on a five-point Likert Scale, with scores ranging from 13 to 65. Higher scores represent higher levels of cancer-related fatigue. For those aged 13 to 18, their fatigue levels will be measured by the Fatigue Scale - Adolescent. It contains 12 items, evaluated on a five-point Likert Scale. Scores range from 12 to 60, and higher scores indicate higher levels of fatigue.
Change in levels of cancer-related fatigue from baseline at 1-month follow-up between intervention and control group | 1-month follow-up
  he Fatigue Scale - Child will be used to assess the fatigue of subjects who are 7 to 12 years old. It contains 13 items, rated on a five-point Likert Scale, with scores ranging from 13 to 65. Higher scores represent higher levels of cancer-related fatigue. For those aged 13 to 18, their fatigue levels will be measured by the Fatigue Scale - Adolescent. It contains 12 items, evaluated on a five-point Likert Scale. Scores range from 12 to 60, and higher scores indicate higher levels of fatigue.
Change in levels of cancer-related fatigue from baseline at 3-month follow-up between intervention and control group | 3-month follow-up
  he Fatigue Scale - Child will be used to assess the fatigue of subjects who are 7 to 12 years old. It contains 13 items, rated on a five-point Likert Scale, with scores ranging from 13 to 65. Higher scores represent higher levels of cancer-related fatigue. For those aged 13 to 18, their fatigue levels will be measured by the Fatigue Scale - Adolescent. It contains 12 items, evaluated on a five-point Likert Scale. Scores range from 12 to 60, and higher scores indicate higher levels of fatigue.
Change in levels of cancer-related fatigue from baseline at 6-month follow-up between intervention and control group | 6-month follow-up
  he Fatigue Scale - Child will be used to assess the fatigue of subjects who are 7 to 12 years old. It contains 13 items, rated on a five-point Likert Scale, with scores ranging from 13 to 65. Higher scores represent higher levels of cancer-related fatigue. For those aged 13 to 18, their fatigue levels will be measured by the Fatigue Scale - Adolescent. It contains 12 items, evaluated on a five-point Likert Scale. Scores range from 12 to 60, and higher scores indicate higher levels of fatigue.
Change in levels of cancer-related fatigue from baseline at 12-month follow-up between intervention and control group | 12-month follow-up
  he Fatigue Scale - Child will be used to assess the fatigue of subjects who are 7 to 12 years old. It contains 13 items, rated on a five-point Likert Scale, with scores ranging from 13 to 65. Higher scores represent higher levels of cancer-related fatigue. For those aged 13 to 18, their fatigue levels will be measured by the Fatigue Scale - Adolescent. It contains 12 items, evaluated on a five-point Likert Scale. Scores range from 12 to 60, and higher scores indicate higher levels of fatigue.
Muscle strength at baseline | Baseline
  Hand-held dynamometer (HHD) will be used to assess the children's right- and left-hand grip strengths.
Change in muscular strength from baseline at 1-month follow-up between intervention and control group | 1-month follow-up
  Hand-held dynamometer (HHD) will be used to assess the children's right- and left-hand grip strengths.
Change in muscular strength from baseline at 3-month follow-up between intervention and control group | 3-month follow-up
  Hand-held dynamometer (HHD) will be used to assess the children's right- and left-hand grip strengths.
Change in muscular strength from baseline at 6-month follow-up between intervention and control group | 6-month follow-up
  Hand-held dynamometer (HHD) will be used to assess the children's right- and left-hand grip strengths.
Change in muscular strength from baseline at 12-month follow-up between intervention and control group | 12-month follow-up
  Hand-held dynamometer (HHD) will be used to assess the children's right- and left-hand grip strengths.
Lung functionality at baseline | Baseline
  A mini-Wright Standard Handheld peak flow meter will be used to determine subjects' peak expiratory flow.
Change in lung functionality from baseline at 1-month follow-up between intervention and control group | 1-month follow-up
  A mini-Wright Standard Handheld peak flow meter will be used to determine subjects' peak expiratory flow.
Change in lung functionality from baseline at 3-month follow-up between intervention and control group | 3-month follow-up
  A mini-Wright Standard Handheld peak flow meter will be used to determine subjects' peak expiratory flow.
Change in lung functionality from baseline at 6-month follow-up between intervention and control group | 6-month follow-up
  A mini-Wright Standard Handheld peak flow meter will be used to determine subjects' peak expiratory flow.
Change in lung functionality from baseline at 12-month follow-up between intervention and control group | 12-month follow-up
  A mini-Wright Standard Handheld peak flow meter will be used to determine subjects' peak expiratory flow.
Quality of life at baseline | Baseline
  The Chinese version of the Pediatric Quality of Life Inventory will be used to measure subjects' quality of life. This scale has 23 items rated on a 5-point Likert scale. These items are categorized into four domains: physical functioning (eight items), emotional functioning (five items), social functioning (five items) and school functioning (five items). The range of possible scores is 0-100, with higher scores representing better quality of Life.
Change in quality of life from baseline at 1-month follow-up between intervention and control group | 1-month follow-up
  The Chinese version of the Pediatric Quality of Life Inventory will be used to measure subjects' quality of life. This scale has 23 items rated on a 5-point Likert scale. These items are categorized into four domains: physical functioning (eight items), emotional functioning (five items), social functioning (five items) and school functioning (five items). The range of possible scores is 0-100, with higher scores representing better quality of Life.
Change in quality of life from baseline at 3-month follow-up between intervention and control group | 3-month follow-up
  The Chinese version of the Pediatric Quality of Life Inventory will be used to measure subjects' quality of life. This scale has 23 items rated on a 5-point Likert scale. These items are categorized into four domains: physical functioning (eight items), emotional functioning (five items), social functioning (five items) and school functioning (five items). The range of possible scores is 0-100, with higher scores representing better quality of Life.
Change in quality of life from baseline at 6-month follow-up between intervention and control group | 6-month follow-up
  The Chinese version of the Pediatric Quality of Life Inventory will be used to measure subjects' quality of life. This scale has 23 items rated on a 5-point Likert scale. These items are categorized into four domains: physical functioning (eight items), emotional functioning (five items), social functioning (five items) and school functioning (five items). The range of possible scores is 0-100, with higher scores representing better quality of Life.
Change in quality of life from baseline at 12-month follow-up between intervention and control group | 12-month follow-up
  The Chinese version of the Pediatric Quality of Life Inventory will be used to measure subjects' quality of life. This scale has 23 items rated on a 5-point Likert scale. These items are categorized into four domains: physical functioning (eight items), emotional functioning (five items), social functioning (five items) and school functioning (five items). The range of possible scores is 0-100, with higher scores representing better quality of Life.

CONTACTS AND LOCATIONS:
Overall Officials: Ho Cheung William Li, Principal Investigator — The University of Hong Kong
Locations (2):
- The University of Hong Kong, Hong Kong, China
- The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cheung AT, Li WHC, Ho LLK, Chan GC, Lam HS, Chung JOK. Efficacy of Mobile Instant Messaging-Delivered Brief Motivational Interviewing for Parents to Promote Physical Activity in Pediatric Cancer Survivors: A Randomized Clinical Trial. JAMA Netw Open. 2022 Jun 1;5(6):e2214600. doi: 10.1001/jamanetworkopen.2022.14600. PMID 35699959